CLINICAL TRIAL: NCT04085380
Title: Identification of New Highly Antibiotic-resistant Bacteria Carriage Risk Factors to Optimize the Detection and Medical Care for Carriers Patients
Brief Title: Digestive Colonisation by Highly Resistant Bacteria (CODBAHRE)
Acronym: CODBAHRE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Other Study IDs: CODBAHRE; APHP180561 (Other: AP-HP); 2019-A01226-51 (Other: IDRCB)
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Risk Factor
Keywords: Clostridium difficile; Multidrug resistant bacteria; Risks factor; highly resistant bacteria; eXDR; ESBL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Rectal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify in hospitalized patients, the risk factors associated with the digestive colonisation by emergent extensively drug-resistant bacteria (eXDR), to optimize their detection and the medical care for carriers these patients

DETAILED DESCRIPTION:
CODBAHRE is a french, regional study, involving 9 centers. Recruitment will take place in all the departments of the centers involved under the supervision of the Infection Control Team.

All patients hospitalized more than 24 hours, on a given day are eligible for the protocol, except the patients unable to answer the questionnaire.

After collecting the non-opposition of the patient, patients will be screened by rectal swab and a questionnaire will be completed.

Each sample will be analyzed to detect eXDR carrying patients.

The carrying patients will be followed during 6 months to estimate the proportion of the population which developped a bacterial infection. This information will be collected by a retrospective telephone survey of carrying patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization of more than 24 hours
* Give his no objection

Exclusion Criteria:

* Hospitalization in psychiatry
* Unwilling to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient hospitalized more than 24 hours, on a given day in one of the participating hospitals, is eligible to be included in the protocol, unless hospitalized in psychiatry
Sampling Method: Non-Probability Sample
Enrollment: 2396 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Risk factors | at inclusion
  Identification of risk factors for digestive colonisation by highly resistant bacteria Lifestyle questionnaire: environment, diet, medical history and result of the rectal swab

SECONDARY OUTCOMES:
Prevalence of multidrug-resistant bacteria will be determined by the number of patients who have been detected at least one multidrug-resistant bacteria referred to the number of patients sampled | 1 day
  Number of patient carrying a Multidrug-resistant bacteria in Ile de France
Prevalence of co-carrying patients of eXDR and ESBL will be determined by the number of patients who carrying eXDR and ESBL referred to the number of patients sampled | 1 day
  Estimate the prevalence of "co-carrying patients of eXDR and ESBL in the Ile de France
Prevalence will be determined by the number of patients who carrying at least one Multidrug-resistant bacteria referred to the number of patients sampled | 1 day
  Establish whether there are significant differences between hospital associated with the recruitment of these institutions.
Proportion of patients carrying "eXDR" who will develop an infection with the same germ referred to the number of eXDR carriers | 6 months
  Estimate the proportion of patients colonized by a "eXDR" who will develop an infection with the same germ.
Cross-transmission rate of eXDR | 1 day
  Number of cross transmissions during the study by comparing the eXDR bacteria genotypes in the same unit
Description of the association between strains (RAPD, infrared Biotyper, genome sequencing). | 16 months
  Identify possible links between strains
Description of resistance and virulence characteristics between strains (RAPD, infrared Biotyper, genome sequencing). | 16 months
  Characterize the resistance and virulence factors of certain strains.
Comparison of the frequency of positive presence of eXDR bacteria obtained between culture technic and molecular biology technic | 16 months
  Comparison culture vs molecular biology technics.

CONTACTS AND LOCATIONS:
Overall Officials: Najiby Kassis-Chikhani, PhD, Principal Investigator — AP-HP, Hôpital Européen Georges Pompidou, Paris; Jean-Ralph Zahar, PhD, Principal Investigator — AP-HP, Hôpitaux Avicenne, Jean Verdier, et René Muret, Bobigny; Véronique Moulin, Principal Investigator — AP-HP, Hôpital Corentin Celton, et Vaugirard; Pierre Frange, PhD, Principal Investigator — AP-HP, Hôpital Necker enfants malades, Paris; Christine Lawrence, PhD, Principal Investigator — AP-HP, Hôpital Raymond Poincaré, Garches; Frédéric Barbut, PhD, Principal Investigator — AP-HP-Hôpital Saint Antoine, Paris
Locations (1):
- HEGP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: one year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization